CLINICAL TRIAL: NCT03401190
Title: An Open-Label, Dose-Response Study of CM4620 Injectable Emulsion (CM4620-IE) in Patients With Acute Pancreatitis and Accompanying Systemic Inflammatory Response Syndrome (SIRS)
Brief Title: CM4620 Injectable Emulsion Versus Supportive Care in Patients With Acute Pancreatitis and SIRS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CalciMedica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CM4620-201
Record Dates: First submitted 2017-12-26; First posted 2018-01-17 (Actual); Results first posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Acute Pancreatitis; Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Pancreatitis; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose Group (Experimental): Phase 1: Cohorts 1 & 2 will consist of 4 female and 4 male patients enrolled concurrently who will be randomized 3:1 to receive CM4620-IE plus standard of care versus standard of care alone. Planned doses for patients who are randomized to receive CM4620-IE are 1.0 mg/kg on Days 1 and 1.4 mg/kg on Days 2-4.
  Interventions: Drug: CM4620 Injectable Emulsion (Low Dose)
- High Dose Group (Experimental): Phase 2: Cohorts 3 & 4 will consist of 8 female and 8 male patients enrolled concurrently who will be randomized 3:1 to receive CM4620-IE plus standard of care versus standard of care alone. Planned doses for patients who are randomized to receive CM4620-IE are 2.08 mg/kg of CM4620-IE on Days 1 and 2, and 1.6 mg/kg on Days 3 and 4.
  Interventions: Drug: CM4620 Injectable Emulsion (High Dose)
- Standard of Care (No Intervention): For all cohorts, patients will be randomized 3:1 to CM4620-IE plus standard of care versus standard of care alone.

INTERVENTIONS:
Drug: CM4620 Injectable Emulsion (Low Dose) — CM4620-IE 1.0 mg/kg on Day 1 and then 1.4 mg/kg on Days 2-4, during the first phase of the study (Cohorts 1 and 2). All doses of CM4620-IE will be administered intravenously (IV) over 4 hours.
  Other Names: CM4620-IE (Low Dose)
  Arms: Low Dose Group
Drug: CM4620 Injectable Emulsion (High Dose) — CM4620-IE 2.08 mg/kg on Days 1 and 2 and then 1.6 mg/kg on Days 3 and 4, during the second phase of the study (Cohorts 3 and 4). All doses of CM4620-IE will be administered intravenously (IV) over 4 hours.
  Other Names: CM4620-IE (High Dose)
  Arms: High Dose Group

SUMMARY:
This open-label, dose-response study will evaluate the safety and efficacy of CM4620-IE in patients with acute pancreatitis and accompanying SIRS. The study will consist of two phases. The first phase will consist of 4 female and 4 male patients (cohorts 1 and 2, respectively), enrolled concurrently, randomized in a 3:1 ratio to receive CM4620-IE plus standard of care versus standard of care alone. Planned doses for first phase will be CM4620-IE 1.0 mg/kg on Day 1 and then 1.4 mg/kg on Days 2 - 4.

The second phase will consist of 8 female and 8 male patients (cohorts 3 and 4, respectively), enrolled concurrently, randomized in a 3:1 ratio to receive CM4620-IE plus standard of care versus standard of care alone. Planned doses for second phase will be CM4620-IE 2.08 mg/kg on Days 1 and 2 and then 1.6 mg/kg on Days 3 and 4. Dose escalation to second phase would only occur if needed for efficacy reasons and if no events suggesting a safety signal would occur with higher dosing.

The study is not powered for the analysis of study data with inferential statisitcs as the primary purpose of the study is to explore what endpoints would be most appropriate for future trials.

DETAILED DESCRIPTION:
After review of the efficacy, tolerability and safety data from cohorts 1 and 2 by the sponsor and the United States Food and Drug Administration, the decision was made to continue the low-dose regimen (CM4620-IE 1.0 mg/kg on Day 1 and then 1.4 mg/kg on Days 2 - 4) in cohort 3. Cohort 4 received the high-dose regimen (CM4620-IE 2.08 mg/kg on Days 1 and 2 and then 1.6 mg/kg on Days 3 and 4) as planned. Efficacy analysis were combined because no dose escalation occurred in cohort 3.

Patients were followed for 90 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of acute pancreatitis established by the presence of abdominal pain consistent with acute pancreatitis and 1 of the following 2 criteria:

   1. Serum lipase and/or serum amylase > 3 times the upper limit of normal (ULN);
   2. Characteristic findings of acute pancreatitis on abdominal imaging;
2. A SpO2 <96% with a FiO2 of 21% (room air) to 27%, or a SpO2 <97% with a FiO2 ≥28%;
3. Diagnosis of SIRS, defined by the presence of at least 2 of the following 4 criteria:

   1. Temperature < 36°C or > 38°C;
   2. Heart rate > 90 beats/minute;
   3. Respiratory rate >20 breaths/minute or arterial carbon dioxide tension (PaCO2) <32 mmHg;
   4. White blood cell count (WBC) >12,000 mm3, or <4,000 mm3, or > 10% immature (band) forms;
4. No evidence of pancreatic necrosis on contrast-enhanced computed tomography (CECT performed in the 18 hours prior to consent or after consent and before Day 1;
5. Adults ≥ 18 years of age;
6. A female patient of child bearing potential who is sexually active with a male partner must be willing to practice acceptable methods of birth control for 365 days after the last dose of CM4620-IE;
7. A male patient who is sexually active with a female partner of childbearing potential must be willing to practice acceptable methods of birth control for 365 days after the last dose of CM4620-IE and must not donate sperm for 365 days.
8. Willing and able to, or have a legal authorized representative (LAR) that is willing and able to, provide informed consent to participate, and to cooperate with all aspects of the protocol.

Exclusion Criteria:

1. Any concurrent clinical condition that a study physician believes could potentially pose an unacceptable health risk to the patient while involved in the study, including a CV SOFA score of 4 at the time of screening, or may limit expected survival to <6 months;
2. Suspected presence of cholangitis in the judgment of the treating investigator;
3. ERCP performed in the previous 7 days;
4. Any malignancy being treated with chemotherapy or immunotherapy;
5. Any autoimmune disease being treated with immunosuppressive medication or immunotherapy;
6. History of:

   1. Acute pancreatitis with pancreatic necrosis on Contrast-Enhanced Computed Tomography (CECT) of the pancreas;
   2. Chronic pancreatitis, pancreatic necrosis or necrosectomy, or pancreatic enzyme replacement therapy;
   3. Biopsy proven cirrhosis, portal hypertension, hepatic failure/hepatic encephalopathy;
   4. Known hepatitis B or C, or HIV;
   5. History of organ or hematologic transplant;
   6. Resuscitated cardiac arrest, myocardial infarction, revascularization, cardiovascular accident (CVA) in the 30 days prior to Day 1;
7. Current renal replacement therapy;
8. Current known abuse of cocaine or methamphetamine;
9. Known to be pregnant or are nursing;
10. Participated in another study of an investigational drug or therapeutic medical device in the 30 days prior to Day 1;
11. History of allergy to eggs or known hypersensitivity to any components of CM4620-IE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Hebbar, MD, Study Director — Chief Medical Officer
Locations (9):
- United States (9):
  - Detroit Receiving Hospital (Wayne State), Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Sinai-Grace Hospital (Wayne State), Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - MetroHealth (Case Western), Cleveland, Ohio
  - Riverside Methodist, Columbus, Ohio
  - Ben Taub (Baylor College of Medicine), Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bruen C, Miller J, Wilburn J, Mackey C, Bollen TL, Stauderman K, Hebbar S. Auxora for the Treatment of Patients With Acute Pancreatitis and Accompanying Systemic Inflammatory Response Syndrome: Clinical Development of a Calcium Release-Activated Calcium Channel Inhibitor. Pancreas. 2021 Apr 1;50(4):537-543. doi: 10.1097/MPA.0000000000001793. PMID 33939666

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Group: Patients were randomized to receive CM4620-IE 1.0 mg/kg on Days 1 and 1.4 mg/kg on Days 2-4. All doses of CM4620-IE were administered intravenously (IV) over 4 hours.
- High Dose Group: Patients were randomized to receive CM4620-IE 2.08 mg/kg on Days 1 and 2, and 1.6 mg/kg on Days 3-4. All doses of CM4620-IE will be administered intravenously (IV) over 4 hours.
- Standard of Care Group: Patients were randomized to receive local standard of care.
Period: Overall Study
Arm/Group | Low Dose Group | High Dose Group | Standard of Care Group
Started | 8 | 6 | 7
Completed | 8 | 4 | 7
Not Completed | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low Dose Group: Consisted of 8 patients, 5 female and 3 male, who were randomized to receive CM4620-IE 1.0 mg/kg on Days 1 and 1.4 mg/kg on Days 2-4. All doses of CM4620-IE were administered intravenously (IV) over 4 hours.
- High Dose Group: Consisted of 6 male patients were randomized to receive CM4620-IE 2.08 mg/kg on Days 1 and 2, and 1.6 mg/kg on Days 3-4. All doses of CM4620-IE will be administered intravenously (IV) over 4 hours.
- Standard of Care Group: Consisted of 7 patients, 4 female and 3 male, who received local standard of care.
- Total: Total of all reporting groups
Arm/Group | Low Dose Group | High Dose Group | Standard of Care Group | Total
Number analyzed (Participants) | 8 | 6 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (14.7) | 44.3 (7.1) | 54.9 (10.7) | 48.1 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 4 | 9
  Male | 3 | 6 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 8 | 4 | 7 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 3 | 6
  White | 6 | 4 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: The Safety and Tolerability of CM4620-IE in Patients With Acute Pancreatitis and Accompanying Systemic Inflammatory Response Syndrome (SIRS) or Hypoxemia.
Description: Safety and tolerability will be assessed by monitoring the frequency, duration and severity of treatment-emergent adverse events (TEAEs) throughout the study period.
Time Frame: 90 Days
Measure: Count of Participants; unit: Participants
Groups:
- Low Dose Group + SC: Consisted of 8 patients, 5 female and 3 male, who were randomized to receive CM4620-IE 1.0 mg/kg on Days 1 and 1.4 mg/kg on Days 2-4. All doses of CM4620-IE were administered intravenously (IV) over 4 hours. All patients were also to receive standard of care (SC).
- High Dose Group + SC: Consisted of 6 male patients were randomized to receive CM4620-IE 2.08 mg/kg on Days 1 and 2, and 1.6 mg/kg on Days 3-4. All doses of CM4620-IE will be administered intravenously (IV) over 4 hours. All patients were also to receive standard of care (SC).
- Standard of Care Group (SC): Consisted of 7 patients, 4 female and 3 male, who received local standard of care.
Arm/Group | Low Dose Group + SC | High Dose Group + SC | Standard of Care Group (SC)
Number analyzed (Participants) | 8 | 6 | 7
Participants
  TEAE patients | 7 | 5 | 3
  Severe TEAE patients | 0 | 2 | 2
  SAE patients | 2 | 1 | 2
  TEAEs leading to discontinuation | 0 | 2 | 0
  TEAEs leading to death | 0 | 1 | 0
  Treatment-related TEAEs | 0 | 1 | 0

2. Secondary Outcome: The Number of Patients With a Change in Computed Tomography Severity Index (CTSI) Score Between Screening and Day 5 (or Discharge, if Earlier)
Description: CTSI score measures abnormal pancreatic morphology and is the sum of two subscales. The Balthazar subscale rates pancreatic CT image findings on a scale of 0 (normal) to 4 (2 or more peri-pancreatic fluid collections. The Pancreatic Necrosis subscale rates pancreatic necrosis from 0 (none) to 6 (>50%). The two subscales are summed for a CTSI score of 0-3 (mild AP), 4-6 (moderate AP), and 7-10 (severe AP).
Time Frame: 5 days (or discharge, if earlier)
Population: One patient treated with the high dose regimen+SC did not receive a CTSI score at either the Screening or Day 5 or Discharge CECTs. One patient treated with SC alone did not receive a CTSI score at Screening because contrast was not given.
Measure: Count of Participants; unit: Participants
Groups:
- High Dose Group + SC: Consisted of 5 male patients were randomized to receive CM4620-IE 2.08 mg/kg on Days 1 and 2, and 1.6 mg/kg on Days 3-4. All doses of CM4620-IE will be administered intravenously (IV) over 4 hours. All patients were also to receive standard of care (SC).
Arm/Group | Low Dose Group + SC | High Dose Group + SC | Standard of Care Group (SC)
Number analyzed (Participants) | 8 | 5 | 7
Participants
  Screening: number analyzed (Participants) | 8 | 5 | 6
  Screening: Number of Patients with Mild AP | 4 | 1 | 2
  Screening: Number of Patients with Moderate AP | 4 | 4 | 3
  Screening: Number of Patients with Severe AP | 0 | 0 | 1
  Day 5 or Discharge, if earlier: Number of Patients with Mild AP | 7 | 1 | 3
  Day 5 or Discharge, if earlier: Number of Patients with Moderate AP | 1 | 4 | 3
  Day 5 or Discharge, if earlier: Number of Patients with Severe AP | 0 | 0 | 1

3. Secondary Outcome: The Number of Patients Tolerating Solid Food
Description: Defined as eating ≥ 50% of a solid meal without vomiting or an increase in pain
Time Frame: at 72 hours (or discharge, if earlier)
Measure: Number; unit: number of patients tolerating solid food
Groups:
- Standard of Care (SC): Consisted of 7 patients, 4 female and 3 male, who received local standard of care.
Arm/Group | Low Dose Group + SC | High Dose Group + SC | Standard of Care (SC)
Number analyzed (Participants) | 8 | 6 | 7
number of patients tolerating solid food | 5 | 2 | 1

4. Secondary Outcome: The Number of Patients Tolerating Solid Food
Description: Defined as eating ≥ 50% of a solid meal without vomiting or an increase in pain
Time Frame: at Day 10 (or discharge, if earlier)
Measure: Number; unit: number of patients tolerating solid food
Arm/Group | Low Dose Group + SC | High Dose Group + SC | Standard of Care (SC)
Number analyzed (Participants) | 8 | 6 | 7
number of patients tolerating solid food | 8 | 5 | 3

5. Secondary Outcome: Percentage of Patients With Persistent Systemic Inflammatory Response Syndrome (SIRS)
Description: The presence of SIRS was defined as the presence of at least 2 of the following 4 criteria:
  * Temperature < 36°C or > 38°C;
  * Heart rate > 90 beats/minute;
  * Respiratory rate > 20 breaths/minute or arterial carbon dioxide tension (PaCO2) < 32 mmHg;
  * White blood cell count (WBC) > 12,000 cells/mm3 or < 4,000 cells/mm3 or > 10% immature (band) forms.
  * The SIRS score was determined at Screening, prior to randomization, and every 12 hours until Day 6, after which it was determined every 24 hours.
Time Frame: ≥ 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Group + SC | High Dose Group + SC | Standard of Care (SC)
Number analyzed (Participants) | 8 | 6 | 7
Participants | 1 | 4 | 5

6. Secondary Outcome: IL-6 Values in Patients With a Maximum IL-6 Value ≥ 150 pg/mL in the First 24 Hours
Description: Assess blood serum samples to be analyzed for interleuken (IL-6) llevels pg/mL collected in the first 24 hours and daily thereafter. Samples were sent to the central laboratory. The results were not provided to the Principal Investigator or treating physician.
Time Frame: Day 10 (or discharge, if earlier)
Population: Only patients with a maximum IL-6 value ≥ 150 pg/mL in the first 24 hours were analyzed. Further, since some patients IL-6 values decreased below 150 pg/mL, they are not displayed in the results table. Analysis only included patients who still had IL-6 values ≥ 150 pg/mL at Day 10 or discharge (whichever was earlier).
Measure: Count of Participants; unit: Participants
Groups:
- Low Dose Group + SC: Consisted of 8 patients, 5 female and 3 male, who were randomized to receive CM4620-IE 1.0 mg/kg on Days 1 and 1.4 mg/kg on Days 2-4. All doses of CM4620-IE were administered intravenously (IV) over 4 hours. All patients also were to receive standard of care (SC).
- High Dose Group + SC: Consisted of 6 male patients were randomized to receive CM4620-IE 2.08 mg/kg on Days 1 and 2, and 1.6 mg/kg on Days 3-4. All doses of CM4620-IE will be administered intravenously (IV) over 4 hours. All patients also were to receive standard of care (SC).
Arm/Group | Low Dose Group + SC | High Dose Group + SC | Standard of Care Group (SC)
Number analyzed (Participants) | 4 | 3 | 3
Participants
  Admission IL-6 Levels: IL-6 ≥ 1000 pg/mL | 0 | 2 | 0
  Admission IL-6 Levels: 150 pg/mL ≤ IL-6 < 1000 pg/mL | 4 | 1 | 3
  Day 10 or discharge IL-6 Levels: number analyzed (Participants) | 0 | 1 | 2
  Day 10 or discharge IL-6 Levels: IL-6 ≥ 1000 pg/mL | 0 | 0 | 0
  Day 10 or discharge IL-6 Levels: 150 pg/mL ≤ IL-6 < 1000 pg/mL | 0 | 1 | 2

7. Secondary Outcome: Median Days in Hospital
Description: Length of stay in hospital in days (randomization to discharge)
Time Frame: discharge
Measure: Median (Full Range); unit: days
Arm/Group | Low Dose Group + SC | High Dose Group + SC | Standard of Care Group (SC)
Number analyzed (Participants) | 8 | 6 | 7
days | 3.06 [1.5 to 8.2] | 6.97 [1.8 to 18.3] | 6.02 [1.1 to 30.0]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 90 days after randomization.
Arm/Group | Low Dose Group | High Dose Group | Standard of Care Group
All-Cause Mortality (participants affected / at risk) | 0/8 | 1/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/8 | 1/6 | 2/7
Other Adverse Events (participants affected / at risk) | 7/8 | 5/6 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Group (N=8) | High Dose Group (N=6) | Standard of Care Group (N=7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cystitis Non-infective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hypoxic-Ischemic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pulseless Electrical Activity (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Group (N=8) | High Dose Group (N=6) | Standard of Care Group (N=7)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Normocytic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Compartment Syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular extra-systoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary dilation (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Scrotal edema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03401190/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT03401190/SAP_001.pdf